CLINICAL TRIAL: NCT01102166
Title: Effect of the Use the Acapella Device in Regional Lung Deposition of Radio-aerosol
Brief Title: Acapella With Nebulization in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Armele Dornelas de Andrade, Universidade Federal de Pernambuco
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: fabricio 01
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: This study was conducted in healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Acapella with nebulization — 1. st Phase In this phase the jet nebulizer was connected to the branch end of the Acapella according to manufacturer's recommendations.
     The volunteer did the radio-aerosol inhalation to obtain images of the lung fields scintigraphy static during the period of 300 seconds using an array of at 256x256x16 incidence later, as that encompasses most incidence of lung volume.
  2. nd Phase The experimental procedure of this phase was similar to the 1st stage, but what differed was it made an adjustment by placing a pipe "T" between the mouthpiece and the device Acapella so that the aerosol would be inhaled not pass through the device.
  Stage 3 This stage was considered phase control since the aerosol inhalation was performed through the mouthpiece connected directly to the nebulizer as is routinely used in clinical practice as illustrated. The procedure of this phase followed the same protocol of previous phases.
  Other Names: - Acapella ® device (DHD Healthcare, wampsville, New York); - Activity standardized 25mCI and after the inhalation chamber were placed on scintigraphy (FORTE of Adac Laboratories)

SUMMARY:
Background:

Devices used to facilitate mucus mobilization have been target of several controversies and mainly a few scientific studies that endorse the use of those equipments. According to the principle of acapella® device, it should be used concomitant with nebulization aiming to optimize its performance in bronchial hygiene.

Aims: To assess the effect of acapella® device application in the radioaerosol regional pulmonary deposition through pulmonary scintigraphy in normal subjects.

Materials and method: 10 health individuals, males and mean age of 24,4 ± 2,2 years participated in this study during the three phases of this research: 1st phase were done with nebulization through acapella® device, attached in the final branch according to manufacturer recommendation; in 2nd phase a ¨T¨tube connector were adapted, being nebulizer attached to the mouthpiece and in 3rd phase nebulization were performance through the mouthpiece as routinely used in aerosoltherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Performed spirometry
* According to the criteria of the Guidelines for Pulmonary Function-2002 published by the official organ of the Brazilian Society of Thoracic

Exclusion Criteria:

* Presence of pulmonary pathology;
* Neurological diseases and body temperature greater than 37 º C during the initial evaluation and during intervention
* Respiratory rate (RR) greater than 35ipm.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Radioaerosol regional pulmonary deposition | One year
  For analysis of lung deposition of radio-aerosol in the different lung areas were delineated regions of interest (ROIs), one for each lung, called the right posterior and left posterior. To analyze this deposition, the lung was divided into regions: upper, middle and bottom, and peripheral, central and intermediate.

SECONDARY OUTCOMES:
Spirometric values | One year
  The procedure was performed with the nose occluded by a nose clip and spirometric data were considered the PFE,FVC and FEV1. We used the protocol of Pereira 3 maneuvers being conducted with an interval between the measurements of one minute. According to the American Thoracic Society, as a criterion for inclusion was considering a variation of less than 0.2 L between the tests and is considered the best of three values.

REFERENCES:
- [Result] Franca EE, Dornelas de Andrade AF, Cabral G, Almeida Filho P, Silva KC, Galindo Filho VC, Marinho PE, Lemos A, Parreira VF. Nebulization associated with bi-level noninvasive ventilation: analysis of pulmonary radioaerosol deposition. Respir Med. 2006 Apr;100(4):721-8. doi: 10.1016/j.rmed.2005.07.012. Epub 2005 Aug 31. PMID 16139491
- [Result] Volsko TA, DiFiore J, Chatburn RL. Performance comparison of two oscillating positive expiratory pressure devices: Acapella versus Flutter. Respir Care. 2003 Feb;48(2):124-30. PMID 12556253
- [Derived] Mesquita FO, Galindo-Filho VC, Neto JL, Galvao AM, Brandao SC, Fink JB, Dornelas-de-Andrade A. Scintigraphic assessment of radio-aerosol pulmonary deposition with the acapella positive expiratory pressure device and various nebulizer configurations. Respir Care. 2014 Mar;59(3):328-33. doi: 10.4187/respcare.02291. Epub 2013 Aug 6. PMID 23920214